CLINICAL TRIAL: NCT03095807
Title: Investigation on Safety, Tolerability and Pharmacokinetics of Single Ascending Doses of NNC9204-1706 in Male Subjects Being Overweight or With Obesity
Brief Title: Investigation of Single Ascending Doses of NNC9204-1706 in Male Subjects Being Overweight or With Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9423-4302; U1111-1177-7821 (Other: World Health Organization (WHO))
Record Dates: First submitted 2017-03-24; First posted 2017-03-30 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NNC9204-1706 A (Experimental)
  Interventions: Drug: NNC9204-1706 A
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNC9204-1706 A — Administered subcutaneously (s.c., under the skin) Up to 7 dose cohorts will be investigated.
  Arms: NNC9204-1706 A
Drug: Placebo — Administered subcutaneously (s.c., under the skin)
  Arms: Placebo

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to assess the safety and tolerability of single doses of NNC9204-1706 administered subcutaneously in male subjects being overweight or with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged 18-55 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between 25.0 and 34.9 kg/m^2 (both inclusive) at screening. Overweight should be due to excess of adipose tissue, as judged by the investigator

Exclusion Criteria:

* Any disorder which in the investigator's opinion might jeopardise subject's safety, evaluation of results, or compliance with the protocol
* Subjects, aged at least 40 years, with an estimated 10-year atherosclerotic cardiovascular disease (ASCVD) (as described in the American College of Cardiology and the American Heart Association Prevention Guideline) risk equal to or above 5%
* Male subjects who are not sexually abstinent or surgically sterilised (vasectomy) and are sexually active with female partner(s) and who are not using a highly effective method of contraception (such as condom with spermicide) combined with a highly effective method of contraception for their non-pregnant female partner(s) (Pearl Index below 1%, such as implants, injectables, oral contraceptives, intrauterine devices, diaphragm or cervical cap+spermicide), and/or intend to donate sperm in the period from screening until 3 months following administration of the investigational medical product

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events (TEAEs) | From the time of dosing (Day 1) and until completion of the post-treatment follow-up visit (Days 10-13)
  Count and % of events

SECONDARY OUTCOMES:
Area under the NNC9204-1706 plasma concentration-time curve | Day 1- Day 7
  Calculated based on NNC9204-1706 measured in blood.
Area under the NNC9204-1706 plasma concentration-time curve (0-24h) | Day 1- Day 7
  Calculated based on NNC9204-1706 measured in blood.
Area under the NNC9204-1706 plasma concentration-time curve (0- to last quantifiable sample) | Day 1- Day 7
  Calculated based on NNC9204-1706 measured in blood.
Maximal observed concentration of the NNC9204-1706 plasma concentration curve | Day 1- Day 7
  Calculated based on NNC9204-1706 measured in blood.
Time to observed maximum concentration of NNC9204-1706 in plasma | Day 1- Day 7
  Calculated based on NNC9204-1706 measured in blood.
Terminal half-life of NNC9204-1706 | Day 1- Day 7
  Calculated based on NNC9204-1706 measured in blood.
Mean residence time of NNC9204-1706 | Day 1- Day 7
  Calculated based on NNC9204-1706 measured in blood.
The apparent total plasma clearance of NNC9204-1706 | Day 1- Day 7
  Calculated based on NNC9204-1706 measured in blood.
The apparent volume of distribution of NNC9204-1706 | Day 1- Day 7
  Calculated based on NNC9204-1706 measured in blood.
Changes in Body weight | Day 1, Days 10-13
  Measured in kg and/or %
Number of injection-site reactions | From the time of dosing (Day 1) to the follow-up visit (Days 10-13)
  Count of reactions
Number of hypoglycaemic episodes | from time of dosing (Day 1) to the follow-up visit (Days 10-13)
  Count of episodes

CONTACTS AND LOCATIONS:
Locations (1):
- Novo Nordisk Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com